CLINICAL TRIAL: NCT00810901
Title: Multimedia Intervention to Motivate Ethnic Teens to be Designated Donors
Brief Title: Intervention to Motivate Teens to be a Designated Organ Donor on Driver's License
Acronym: Idecide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK079684; R01DK079684 (NIH); R01DK079684-03S1 (NIH)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-01

CONDITIONS: Tissue and Organ Procurement; Alcohol Abstinence
Keywords: ethnic minority adolescents; designated organ donor
MeSH Terms: conditions — Alcohol Abstinence | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Organ Donor (Experimental): Intervention used a DVD, text messaging, emails, a website, US Mail, and telephone calls to educate teens about their choice to become a designated organ donor on their first driver's license application.
  Interventions: Behavioral: Organ Donor
- Alcohol Prevention (Active Comparator): Intervention used a DVD and text messages, to educate teens about the laws that prohibit underage minors purchasing and consuming alcohol
  Interventions: Behavioral: Alcohol Prevention

INTERVENTIONS:
Behavioral: Organ Donor — Subjects receive information about becoming a designated organ donor -via DVD, email, text messaging, website, and US mail.
  Other Names: Idecide Project
  Arms: Organ Donor
Behavioral: Alcohol Prevention — Use DVD, website, text messaging, email and US mail to educate teenagers about the consequences associated with purchasing and using alcohol.
  Other Names: Roll of the Dice
  Arms: Alcohol Prevention

SUMMARY:
This study will test the effectiveness of a multimedia campaign to educate ethnic minority teens about the choice to become a designated organ donor on their first driver's license.

DETAILED DESCRIPTION:
Less than a fourth of ethnic minority teens in the U.S. are a designated donor (DD) on their state-issued driver's license. Asian-American/Pacific Islander (AA/PI) adolescents in Hawaii are even less likely to be a DD or to have talked to their family about becoming an organ donor. Health education interventions for adolescents have demonstrated improvements in knowledge and intentions to be an organ donor; but, AA/PI teens are underrepresented in such studies. Nevertheless, whether changes in knowledge or intentions result in more organ donors is unclear, since previous studies have not included a concrete behavioral outcome such as the teen becoming a donor on their driver's license. This application will test, via a randomized clinical trial, the efficacy of an Interactive Multimedia Intervention (IMI) to increase the number of AA/PI adolescents who are a DD on their state issued driver's license, identification card, or organ donor card/donor registry. Teen groups will be recruited from the community (churches and high schools, n = 40 groups, 530 teens) and randomly assigned to either the intervention or a comparison condition on prevention of underage drinking of alcohol. The theoretically-derived intervention will include culturally sensitive messages and information about being a designated donor that will be delivered via a DVD, Email, text/instant messaging, and websites. The comparison condition includes materials (DVD) previously shown to increase awareness about laws restricting access to alcohol by teens. The primary outcome is objectively validated donor status on a teens' driver's license/state identification card (ID) or donor card after 12 months of intervention. A secondary outcome is the reported rate of family discussions about organ donation and knowledge/intentions about donation. We hypothesize the youth groups assigned to the intervention will have higher rates for family discussions and DD status, compared to groups in the comparison condition. We will also test whether psychosocial and cultural factors act as mediators of any change in teens' knowledge, attitudes & stages of change to become a DD. After the randomized trial we will disseminate the intervention to Organ Procurement Organizations in Hawaii and other states, and track diffusion outcomes over a year. If IMI methods can increase the number of minority teens who become a DD on their driver's license by 10% this would translate to 500,000 more teenage designated donors in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* adolescent aged 14-19
* member of a school club, youth program or teen group
* read and speak English
* parent provides consent

Exclusion Criteria:

* plans to permanently move out of state

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 429 (Actual)
Dates: Start 2008-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Albright, PhD, MPH, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii School of Nursing and Dental Hygiene, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Organ Donor: Intervention used a digital video disk (DVD), text messaging, emails, a website, US Mail, and telephone calls to educate teens about their choice to become a designated organ donor on their first driver's license application.
  Organ Donor: Subjects receive information about becoming a designated organ donor -via DVD, email, text messaging, website, and US mail.
- Alcohol Prevention: Intervention used a digital video disk (DVD) and text messages, to educate teens about the laws that prohibit underage minors purchasing and consuming alcohol
  Alcohol Prevention: Use DVD, website, text messaging, email and US mail to educate teenagers about the consequences associated with purchasing and using alcohol.
Period: Overall Study
Arm/Group | Organ Donor | Alcohol Prevention
Started | 253 | 176
1-month Follow up | 242 | 146
6-month Follow-up | 181 | 122
Completed | 165 | 118
Not Completed | 88 | 58
Not completed — Lost to Follow-up | 88 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Organ Donor | Alcohol Prevention | Total
Number analyzed (Participants) | 253 | 176 | 429
Age, Continuous [Mean (Standard Deviation); unit: years] — mean age by study condition
  years | 15.8 (1.2) | 16.1 (1.3) | 15.9 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 87 | 213
  Male | 127 | 89 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 35 | 68
  Not Hispanic or Latino | 209 | 130 | 339
  Unknown or Not Reported | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 147 | 95 | 242
  Native Hawaiian or Other Pacific Islander | 50 | 46 | 96
  Black or African American | 0 | 3 | 3
  White | 21 | 15 | 36
  More than one race | 35 | 16 | 51
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 253 | 176 | 429
Designated organ donor on driver's license [Number; unit: participants]
  Organ donor on license at baseline | 52 | 39 | 91
  Not organ donor on license at baseline | 201 | 137 | 338

OUTCOME MEASURES:

1. Primary Outcome: Designated Organ Donor Status on Driver's License
Description: Number of students who reported not being donor at baseline but were donor at 12 months follow-up
Time Frame: 12 months
Population: t-test
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Alcohol Prevention | Organ Donor
Number analyzed (Participants) | 118 | 165
participants | 67 [63 to 71] | 38 [36 to 40]

2. Secondary Outcome: Talked to Parents About Choice to be Organ Donor on License at 12 Months
Description: Number of teens who talk had not talked to parents at baseline but reported they had talked to their parents about the choice to become an organ donor on their driver's license at 12 months
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Alcohol Prevention | Organ Donor
Number analyzed (Participants) | 118 | 165
participants | 80 [73 to 87] | 74 [63 to 85]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Alcohol Prevention | Organ Donor
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/176
Other Adverse Events (participants affected / at risk) | 3/253 | 2/176
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcohol Prevention (N=253) | Organ Donor (N=176)
Emotional reaction (Social circumstances) | 3 (3) | 2 (2) — Student became upset about condition-specific issue (i.e,. underage drinking problem) or had argument with parent about condition-specific issue (i.e., becoming organ donor on driver's license)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No